CLINICAL TRIAL: NCT04683198
Title: A Single -Arm, Open-label, Multicenter Phase II Study of Camrelizumab Combined With Apatinib ,Carboplatin and Etoposide in Participants With Untreated Extensive-Stage (ES) Small Cell Lung Cancer (SCLC)
Brief Title: Camrelizumab Combined With Apatinib ,Carboplatin and Etoposide in Participants With ES-SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-SCLC-II-001
Record Dates: First submitted 2020-12-17; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-10

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — camrelizumab; apatinib; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: camrelizumab +apatinib+ Carboplatin + Etoposide (Experimental): Induced stage：camrelizumab 200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Apatinib capsules 250 mg given orally +Etoposide (100mg/m2 IV continuously on Day 1, 2 and 3）+Carboplatin（AUC 5 mg/mL/min IV on Day 1 ; maintenance stage：Camrelizumab 200 mg administered intravenously (IV) on Day 1 of each 21-day cycle plus Apatinib capsules 250 mg given orally, once daily in 21-day cycle .
  Interventions: Drug: camrelizumab; Drug: Apatinib Mesylate; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: camrelizumab — Camrelizumab intravenous infusion was administered at a dose of 200 mg on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4/6) and maintenance phase ,until PD.
  Other Names: SHR-1210
Drug: Apatinib Mesylate — Apatinib capsules 250 mg given orally , once daily in 21-day cycle and maintenance phase,until PD.
Drug: Carboplatin — Carboplatin intravenous infusion to achieve an initial target AUC of 5 mg/mL/min was administered on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4/6).
Drug: Etoposide — Etoposide intravenous infusion was administered at a dose of 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle during the induction phase (Cycles 1-4/6).

SUMMARY:
This single-arm, Phase II, multicenter study was designed to evaluate the safety and efficacy of Camrelizumab (anti-programmed death-receptor 1 [PD-1] antibody) in combination with Apatinib+carboplatin plus (+) etoposide in chemotherapy-naive participants with ES-SCLC. Participants will be receive camrelizumab +apatinib+ carboplatin + etoposide on 21-day cycles for four -six cycles in the induction phase followed by maintenance with camrelizuab +apatinib until progressive disease (PD) as assessed by the investigator using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). Treatment can be continued until persistent radiographic PD or symptomatic deterioration.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 70 years old
* Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system);
* No prior systemic treatment for ES-SCLC；
* Has received radiotherapy and chemotherapy for limited stage SCLC must have received definitive treatment, and has at least 6 months of no treatment interval from the last treatment to the diagnosis of extensive SCLC
* Eastern Cooperative Oncology Group performance status of 0 or 1；
* life expectancy≥ 12 weeks
* Adequate hematologic and organ function
* Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study (such as intrauterine devices , contraceptives or condoms) ; No pregnant or breastfeeding women, and a negative pregnancy test are received within 72h before the first dose of the study.

Exclusion Criteria:

* Has prior therapy with apatinib,anlotinib, anti-programmed cell death (PD)-1, anti-PD-L1 or other immunotherapy against PD-1/PD-L1;
* Has active or untreated central nervous system (CNS) metastases and/or cancerous meningitis;
* Has spinal cord compression which was not cured or relieved through surgery and/or radiotherapy, or diagnosed spinal cord compression after treatment showed no clinical evidence of disease stabilization prior to allocation ≥1 week;
* Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary with blood vessels is unclear;
* Active autoimmune diseases requiring systemic treatment occurred within 2 years prior to first administration ;
* Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10 mg/day prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first administration;
* Has arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident including transient ischemic attack, deep vein thrombosis and pulmonary embolism;
* Within 3 months prior to initial administration, subjects with evidence of bleeding had clinical significance or history of bleeding tendency, regardless of severity;
* Has vaccinated with vaccines or attenuated vaccines within 4 weeks prior to first administration
* Has major surgical procedure、biopsy or obvious traumatic injury within 28 days before allocation;
* Has participated in other anticancer drug clinical trials within 4 weeks;
* Has diagnosed and/or treated additional malignancy within 5 years prior to allocation. Exceptions include cured basal cell carcinoma of skin and carcinoma in situ of cervix;
* Has any severe and/or uncontrolled disease;
* Has adverse events caused by previous therapy except alopecia that did not recover to ≤ grade 1;
* Has drug abuse history that unable to abstain from or mental disorders; 13. Has any severe and/or uncontrolled disease;
* Severe hypersensitivity occurs after administration of other monoclonal antibodies;
* According to the judgement of the researchers, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed by the Investigator Using RECIST v1.1 | Baseline until PD or death, whichever occurs first (up to approximately 13 months)
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least 20% increase in the sum of the longest diameter of target lesions compared to baseline, or unequivocal progression in non-target lesion(s), or the appearance of new lesion(s).

SECONDARY OUTCOMES:
Overall survival (OS) | up to approximately 20 months
  Baseline until death from any cause
Overall response rate (ORR) | up to 12 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) .
Disease control rate (DCR) | up to 12 months
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Duration of response（DOR） | up to 12 months
  For participants who demonstrate CR or PR, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first
PFS rate of 6 months progression-free survival | up to 6 months
  PFS rate of progression-free survival at 6 months: the percentage of subjects who did not develop disease progression or die of any cause at 6 months after beganing.

IPD SHARING:
Plan to Share IPD: No